CLINICAL TRIAL: NCT03293238
Title: Practical Indications for Sonography in Musculoskeletal Medicine-Knee Joint Injections
Brief Title: Ultrasound Guided Knee Injections in Musculoskeletal Medicine
Acronym: PRISMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrews Research & Education Foundation (Other)
Collaborators: American Medical Society for Sports Medicine (AMSSM) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRISMM-Knee
Record Dates: First submitted 2017-09-18; First posted 2017-09-26 (Actual); Results first posted 2019-11-06 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Knee Osteoarthritis
Keywords: knee; osteoarthritis; ultrasound; sonography; injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of four intervention arms for the purpose of obtaining patient reported outcomes as it relates to the accuracy of injections into the knee joint with or without ultrasound guidance.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blindfolded for the duration of their procedure. Investigator will always place ultrasound probe on patient's knee regardless of group assignment to eliminate bias. To further enhance blinding, the ultrasound screen will placed on freeze for the patients randomized into the groups without ultrasound guidance. Radiologist will be blinded to patient's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Joint Line Ultrasound (Active Comparator): Patients assigned to this group receive a standard medial or lateral joint line injection of Euflexxa aided by ultrasound guidance while sitting up.
  Interventions: Procedure: Joint line ultrasound
- Joint Line Landmark (Sham Comparator): Patients assigned to this group receive a standard medial or lateral joint line injection of Euflexxa without ultrasound guidance while sitting up.
  Interventions: Procedure: Joint line landmark
- Suprapatellar Ultrasound Guided (Active Comparator): Patients assigned to this group receive an injection of Euflexxa while lying down into the suprapatellar pouch aided by ultrasound guidance.
  Interventions: Procedure: Suprapatellar ultrasound guided
- Suprapatellar Landmark (Sham Comparator): Patients assigned to this group receive an injection of Euflexxa while lying down into the suprapatellar pouch without ultrasound guidance.
  Interventions: Procedure: Suprapatellar Landmark

INTERVENTIONS:
Procedure: Joint line ultrasound — Patients will be sitting with knee bent at 90 degrees. Clinician will palpate extremity to determine if a medial or lateral approach will be made for the injection of Euflexxa into the joint space. The procedure will be aided by real time visualization utilizing ultrasound guidance.
  Other Names: JLUS
  Arms: Joint Line Ultrasound
Procedure: Joint line landmark — Patients will be sitting with knee bent at 90 degrees. Clinician will palpate extremity to determine if a medial or lateral approach will be made for the injection of Euflexxa into the joint space. The procedure will not be aided by ultrasound guidance, but completed based strictly on tactile feedback from the injecting physician.
  Other Names: JLL
  Arms: Joint Line Landmark
Procedure: Suprapatellar ultrasound guided — Patients will be lying supine on exam table. Ultrasound will be used to capture a longitudinal view of the proximal patella and the plane between the prefemoral fat pad and suprapatellar fat pad. After the desired visualization is achieved, injection of Euflexxa will be made within the suprapatellar pouch.
  Other Names: SPUS
  Arms: Suprapatellar Ultrasound Guided
Procedure: Suprapatellar Landmark — Patients will be lying supine on exam table. Injecting physician will insert needle lateral to the vastus lateralis toward the suprapatellar pouch, and will inject of Euflexxa once it is believed that the needle tip is in the pouch.
  Other Names: SPL
  Arms: Suprapatellar Landmark

SUMMARY:
This study will compare the accuracy and patient reported outcomes between four different techniques used to perform a knee injection.

DETAILED DESCRIPTION:
This study will compare the accuracy and patient-oriented outcomes between various techniques for intra-articular knee injections. Historically, a joint line (intercondylar) technique of injection at the medial or lateral joint line, reliant solely upon clinical palpation, has been the most popular approach among primary care and orthopedic providers. Newer approaches, making use of ultrasound visualization to accomplish access to the intercondylar recess and the anterolateral suprapatellar pouch, have gained in popularity. Because of uncertain accuracy with the traditional approach, this study is designed to determine if sonographic visualization combined with either of these two newer techniques improves accuracy and affects patient-oriented outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 to 90
* Clinician determined need for intra-articular knee injection
* Radiograph confirmed grade 1-4 Kellgren Lawrence osteoarthritis scale

Exclusion Criteria:

* Allergy to contrast dye, shellfish
* Allergy to egg product or hyaluronate
* Allergy to lidocaine
* Localized skin infection at planned site of injection
* Inability to complete follow-up phone call three months following the injection
* Viscosupplementation injection within 6 months of the current evaluation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-11-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Hackel, MD, Principal Investigator — Andrews Institute for Orthopaedic & Sports Medicine
Locations (1):
- Andrews Research & Education Foundation, Gulf Breeze, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peat G, McCarney R, Croft P. Knee pain and osteoarthritis in older adults: a review of community burden and current use of primary health care. Ann Rheum Dis. 2001 Feb;60(2):91-7. doi: 10.1136/ard.60.2.91. PMID 11156538
- [Background] Jackson DW, Evans NA, Thomas BM. Accuracy of needle placement into the intra-articular space of the knee. J Bone Joint Surg Am. 2002 Sep;84(9):1522-7. doi: 10.2106/00004623-200209000-00003. PMID 12208907
- [Background] Wiler JL, Costantino TG, Filippone L, Satz W. Comparison of ultrasound-guided and standard landmark techniques for knee arthrocentesis. J Emerg Med. 2010 Jul;39(1):76-82. doi: 10.1016/j.jemermed.2008.05.012. Epub 2008 Dec 5. PMID 19062223
- [Background] Esenyel C, Demirhan M, Esenyel M, Sonmez M, Kahraman S, Senel B, Ozdes T. Comparison of four different intra-articular injection sites in the knee: a cadaver study. Knee Surg Sports Traumatol Arthrosc. 2007 May;15(5):573-7. doi: 10.1007/s00167-006-0231-6. Epub 2006 Dec 6. PMID 17149645
- [Background] Naredo E, Cabero F, Beneyto P, Cruz A, Mondejar B, Uson J, Palop MJ, Crespo M. A randomized comparative study of short term response to blind injection versus sonographic-guided injection of local corticosteroids in patients with painful shoulder. J Rheumatol. 2004 Feb;31(2):308-14. PMID 14760802
- [Background] Berkoff DJ, Miller LE, Block JE. Clinical utility of ultrasound guidance for intra-articular knee injections: a review. Clin Interv Aging. 2012;7:89-95. doi: 10.2147/CIA.S29265. Epub 2012 Mar 20. PMID 22500117
- [Background] Cunnington J, Marshall N, Hide G, Bracewell C, Isaacs J, Platt P, Kane D. A randomized, double-blind, controlled study of ultrasound-guided corticosteroid injection into the joint of patients with inflammatory arthritis. Arthritis Rheum. 2010 Jul;62(7):1862-9. doi: 10.1002/art.27448. PMID 20222114
- [Background] Im SH, Lee SC, Park YB, Cho SR, Kim JC. Feasibility of sonography for intra-articular injections in the knee through a medial patellar portal. J Ultrasound Med. 2009 Nov;28(11):1465-70. doi: 10.7863/jum.2009.28.11.1465. PMID 19854960
- [Background] Hong BY, Lim SH, Cho YR, Kim HW, Ko YJ, Han SH, Lee JI. Detection of knee effusion by ultrasonography. Am J Phys Med Rehabil. 2010 Sep;89(9):715-21. doi: 10.1097/PHM.0b013e3181e29c55. PMID 20531157

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited through individual physician practices.
Pre-assignment Details: Sixty-three patients were enrolled and randomized into four groups: Group 1: Joint Line Ultrasound Guided (n= 19), Group 2: Joint Line Landmark Based (sham Ultrasound) (n= 16), Group 3: Suprapatellar Ultrasound Guided (n= 14), Group 4: Suprapatellar Landmark Based (sham Ultrasound) (n= 14). One patient's radiographic imaging was lost.
Groups:
- Joint Line Ultrasound: Patients assigned to this group received a standard medial or lateral joint line injection of Euflexxa aided by ultrasound guidance while sitting up.
  Joint line ultrasound: Patients were sitting with knee bent at 90 degrees. Clinician palpated the extremity to determine if a medial or lateral approach would be made for the injection of Euflexxa into the joint space. The procedure was aided by real time visualization utilizing ultrasound guidance.
- Joint Line Landmark: Patients assigned to this group received a standard medial or lateral joint line injection of Euflexxa without ultrasound guidance while sitting up.
  Joint line landmark: Patients were sitting with knee bent at 90 degrees. Clinician palpated the extremity to determine if a medial or lateral approach would be made for the injection of Euflexxa into the joint space. The procedure was not be aided by ultrasound guidance, but completed based strictly on tactile feedback from the injecting physician.
- Suprapatellar Ultrasound Guided: Patients assigned to this group received an injection of Euflexxa while lying down into the suprapatellar pouch aided by ultrasound guidance.
  Suprapatellar ultrasound guided: Patients were lying supine on exam table. Ultrasound was used to capture a longitudinal view of the proximal patella and the plane between the prefemoral fat pad and suprapatellar fat pad. After the desired visualization is achieved, injection of Euflexxa was made within the suprapatellar pouch.
- Suprapatellar Landmark: Patients assigned to this group received an injection of Euflexxa while lying down into the supratpatellar pouch without ultrasound guidance.
  Suprapatellar Landmark: Patients were lying supine on exam table. Injecting physician inserted a needle lateral to the vastus lateralis toward the suprapatellar pouch, and injected of Euflexxa once it is believed that the needle tip is in the pouch.
Period: Overall Study
Arm/Group | Joint Line Ultrasound | Joint Line Landmark | Suprapatellar Ultrasound Guided | Suprapatellar Landmark
Started | 19 | 16 | 14 | 14
Completed | 19 | 16 | 14 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Joint Line Ultrasound | Joint Line Landmark | Suprapatellar Ultrasound Guided | Suprapatellar Landmark | Total
Number analyzed (Participants) | 19 | 16 | 14 | 14 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (12.2) | 65.3 (12.1) | 71.4 (9.6) | 68.8 (9.5) | 67.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 12 | 8 | 41
  Male | 7 | 7 | 2 | 6 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19 | 16 | 14 | 14 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Knee Injection
Description: To assess presence or absence of contrast medium within the target knee joint as determined by a blinded radiologist. If contrast medium could be observed in the joint then the injection was considered a success.
Time Frame: Procedure visit 3 (3-4 weeks after 1st injection)
Population: Number of patients in each group with successful injections into the knee joint.
Measure: Count of Participants; unit: Participants
Arm/Group | Joint Line Ultrasound | Joint Line Landmark | Suprapatellar Ultrasound Guided | Suprapatellar Landmark
Number analyzed (Participants) | 19 | 16 | 14 | 14
Participants | 17 | 14 | 13 | 7

2. Secondary Outcome: Procedural Satisfaction Score at 3 Months Post Injection
Description: Patient reported procedural satisfaction score on scale of 0 to 10. A score of 10 indicates high satisfaction with the procedure.
Time Frame: 3 month follow-up appointment following 3rd injection
Population: ANOVA
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Joint Line Ultrasound | Joint Line Landmark | Suprapatellar Ultrasound Guided | Suprapatellar Landmark
Number analyzed (Participants) | 19 | 16 | 14 | 14
units on a scale | 7.84 (3.13) | 8.71 (2.20) | 7.14 (3.33) | 8.29 (2.76)
Statistical Analysis 1: Comparison: Joint Line Ultrasound vs Joint Line Landmark vs Suprapatellar Ultrasound Guided vs Suprapatellar Landmark; Test type: Superiority; p = 0.527, ANOVA

3. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Score
Description: Compare the Western Ontario and McMaster Universities Osteoarthritis Index between groups at the 3-month follow-up appointment. The scale is 0-100. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Time Frame: Pre-Injection and 3 month follow-up appointment following 3rd injection
Population: Mean WOMAC score Pre-Injection and at 3-months post injection.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Joint Line Ultrasound | Joint Line Landmark | Suprapatellar Ultrasound Guided | Suprapatellar Landmark
Number analyzed (Participants) | 19 | 16 | 14 | 14
units on a scale
  Pre-Injection | 48.05 (30.92) | 43.75 (27.53) | 53.15 (25.25) | 47.61 (30.71)
  Post-Injection | 23.42 (25.88) | 31.07 (28.63) | 32.5 (27.02) | 28.57 (20.70)
Statistical Analysis 1: Comparison: Joint Line Ultrasound vs Joint Line Landmark vs Suprapatellar Ultrasound Guided vs Suprapatellar Landmark; Test type: Superiority; p = 0.749, ANOVA

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Joint Line Ultrasound | Joint Line Landmark | Suprapatellar Ultrasound Guided | Suprapatellar Landmark
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/16 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/16 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/19 | 0/16 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-11-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT03293238/Prot_SAP_000.pdf